CLINICAL TRIAL: NCT03043027
Title: Efficacy of Liposomal Bupivacaine for Pain Control After Percutaneous Nephrostolithotomy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: cost of medicine too expensive to continue without funding
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, David Hoenig, Principal Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB# 16-748
Record Dates: First submitted 2017-01-20; First posted 2017-02-03 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Renal Calculi; Postoperative Pain
MeSH Terms: conditions — Kidney Calculi; Pain, Postoperative | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Liposomal bupivicaine (Experimental)
  Interventions: Drug: liposomal bupivicaine
- bupivicaine (Active Comparator)
  Interventions: Drug: Bupivacaine
- saline (Placebo Comparator)
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: liposomal bupivicaine — local anesthetic
  Arms: Liposomal bupivicaine
Drug: Bupivacaine — local anesthetic
  Arms: bupivicaine
Drug: Saline Solution — saline injection
  Arms: saline

SUMMARY:
Percutaneous nephrostolithotomy (PCNL) is a common endoscopic procedure performed for upper urinary tract calculus disease. Despite being minimally invasive, it is associated with significant postoperative pain, often necessitating inpatient hospitalization and narcotic pain medications. Additionally, one of a number of catheters is often left protruding from the access tract for a period of time following the procedure, adding to patient discomfort. Attempts have been made to study peri-tubular or access tract analgesic installation, which have shown promise.1-2 However, no studies, to our knowledge, have examined the use of liposomal bupivacaine preparations in this regard. In this study we hope to prospectively analyze the use of liposomal bupivacaine injected to the access tract site at the time of PCNL and determine its effects on postoperative narcotic requirement and pain scores.

Patients presenting for PCNL will be randomized to either the liposomal bupivacaine or usual care, which involves no injection of local anesthesia. Patients will then be followed during their inpatient stay. Total narcotic requirement (in milligrams) and pain scores (using Wong-Baker FACES rating scale) will be compared.3 Typical postoperative care and discharge criteria will not change during the course of this study.

DETAILED DESCRIPTION:
Subjects will be randomly assigned by a 1:1:1 ratio to one of the following groups:

1. Saline (control arm)
2. Liposomal bupivicaine (long-acting local anesthetic)
3. Bupivacaine (local anesthetic)

   The Biostatistics Unit will develop a randomization procedure using a permuted block design. Randomization will be stratified by site (LIJ or NSUH). The randomization process will occur in REDCap using the Randomization Module. Details of the procedure, including required record keeping, will be further developed upon approval of this protocol.

   Patients undergoing PCNL will need no alterations of procedure in regards to positioning, obtaining access, or removal of calculi. Efforts will be made to remove the calculus with use of one access tract only; however, if the surgeon performing the procedures deems that additional access tracts are needed they can be obtained. Similarly, efforts will be taken to include a single nephrostomy tube without the need for a ureteral stent. However, if the attending surgeon deems either of these factors need to be altered, he may do so at his discretion. The use of multiple access tracts, multiple nephrostomy tubes, or a ureteral stent will then disqualify the patient from the trial and they shall then be withdrawn from the study. Because of the nature of the procedure, it is difficult to predict with certainty if patients will need any of these alterations and thus these decisions may need to be made intraoperatively.

   If the patient still meets inclusion criteria, 20 mL of agent will be infiltrated subcutaneously depending on what arm the patient was randomized to. 10 mL will be place at the lateral edge of the tract while 10 mL will be placed at the medial edge. The patient will be awakened without any other changes to standard PCNL protocol. All PCNL procedures will be performed in the aforementioned manner by one of three fellowship trained endourologists with high-volume stone practices (David Hoenig, Zeph Okeke, and Arthur Smith).

   The primary outcome being assessed is the patient's pain rating at 24 hours after the procedure. All patient scores will be recorded using a specific VAS, the Wong-Baker FACES Pain Rating Scale. These values will be converted to a numerical scale from 0-10 accordingly. Patients will be assigned a pain rating handout which will be present in their hospital room for 48 hours or until they are discharged, whichever comes first. Nursing staff or a urology inpatient team member will prompt the patient at the 24 hour period to describe their pain using the FACES scale and they will record this on their handout. Nursing or a urology inpatient team member will collect handouts at time of discharge or after 48 hours, whichever comes first.

   Primary Objective:

   To determine the effects of liposomal bupivacaine injections at the access site during PCNL on postoperative pain and narcotic requirement.

   Primary Outcome:

   • Visual analog scale (VAS) at 24 hours (Liposomal bupivicaine vs. bupivicaine only)

   Secondary Outcomes:
   * Total dose of narcotics (mg) over the course of hospital stay
   * VAS pain scores (across time)
   * Length of Stay (LOS)
   * Time-to-first rescue pain medication after surgery

   Randomization:

   Subjects will be randomly assigned by a 1:1:1 ratio to one of the following groups:
4. Saline (control arm)
5. Liposomal bupivicaine (long-acting)
6. Bupivacaine (local anesthetic)

The Biostatistics Unit will develop a randomization procedure using a permuted block design. Randomization will be stratified by site (LIJ or NSUH). The randomization process will occur in REDCap using the Randomization Module. Details of the procedure, including required record keeping, will be further developed upon approval of this protocol.

Statistical Methods:

Descriptive statistics (means ± standard deviations or medians and interquartile range [25th percentile, 75th percentile] for continuous data; frequencies and percentages for categorical data) will be calculated by group.

Comparability of the three groups at baseline will be analyzed using the chi-square test or Fisher's exact test, as deemed appropriate, for categorical variables. Continuous variables such as age and narcotic usage will be compared using Analysis of Variance (ANOVA) or the Kruskal-Wallis test as indicated.

For the primary outcome, the 24 hour VAS score will be compared between the liposomal bupivacaine vs. bupivacaine groups using the two-sample t-test or Mann-Whitney test as deemed appropriate.

A repeated measures analysis of variance (RMANOVA) with a mixed models approach will be used to determine if the groups' trajectories for VAS differ across time, measured at 6, 12, 24, and 48 hours post-operatively (i.e., the group x time interaction). The standard assumptions of Gaussian residuals and equality of variance will be tested. If the normality assumption is not met, a transformation will be used for the analysis of VAS. The repeated within subjects factor will be time and the within subjects factor will be group (Saline, Liposomal bupivicaine, or Bupivacaine).

"Time-to-first rescue pain medication after surgery" will be analyzed by applying standard methods of survival analysis, i.e., computing the Kaplan-Meier product limit curves, where group will be the stratification variable. In cases where the endpoint event, "first rescue pain medication after surgery", did not occur, the number of hours until last follow-up will be used and considered 'censored'. The groups will be compared using the log-rank test. The median "time to first rescue pain medication after surgery" and corresponding 95% confidence intervals for each group will be obtained from the Kaplan-Meier/Product-Limit Estimates.

LOS will also be analyzed using the standard methods of survival described above, however, without any censored data.

A result will be considered statistically significant at the p<0.05 level of significance. Upon finding a significant difference among the three groups in any of the above analyses, Bonferroni adjusted multiple pairwise comparisons will be carried out in order to determine specifically which groups differed from one another. A pairwise comparison will be considered statistically significant if p<0.0167 (=0.05/3).

All analyses will be performed using SAS version 9.4 (SAS Institute Inc., Cary, NC).

Intention-to-Treat (ITT):

Statistical analysis will be performed using the modified intention-to-treat population (mITT), defined as all randomized subjects who receive treatment and who have completed at least one pain score after baseline assessment.

Interim Analysis and Early Stopping:

There are no plans for interim analysis for efficacy.

Sample Size Considerations:

The proposed sample size for this prospective, single-blinded randomized trial is 99 subjects (n=33 per group). The sample size is based on the primary analysis of VAS at 24 weeks between the Liposomal bupivicaine vs. bupivicaine groups. Although other analyses will be performed on all 3 groups, the sample size calculation has been simplified to the analysis of Liposomal bupivicaine vs. bupivicaine at a single time point.

Based on data published by Kirac et al. (2013), the mean 24-hour VAS score for the bupivicaine group was 2.8 ± 0.9. We assume that the VAS score at 24-hours for the Liposomal bupivicaine group will be 25% greater (VAS=3.5). A sample size of 33 in each group will have 80% power to detect such a difference in means of -0.7 assuming that the common standard deviation is 1.0 using a two group t-test with a 0.05 two-sided significance level. Expanding this to 3 groups will yield a total sample size of 99 subjects.

Outcomes The primary outcome being assessed is the patient's pain rating at 24 hours after the procedure. All patient scores will be recorded using a specific VAS, the Wong-Baker FACES Pain Rating Scale. These values will be converted to a numerical scale from 0-10 accordingly. Patients will be assigned a pain rating handout which will be present in their hospital room for 48 hours or until they are discharged, whichever comes first. Nursing staff or a urology inpatient team member will prompt the patient at the 24 hour period to describe their pain using the FACES scale and they will record this on their handout. Nursing or a urology inpatient team member will collect handouts at time of discharge or after 48 hours, whichever comes first.

The following data will also be recorded and serve as the secondary outcomes:

1. Patient's pain rating at 6, 12, and 48 hours in all arms
2. Patient's pain rating at 24 hours in the saline arm
3. Patient length of stay (LOS)
4. Time-to-first rescue pain medication after surgery
5. Total narcotic use
6. Weight adjusted total narcotics use
7. Narcotic density (mg of morphine equivalent/hours) used at 0-6 hours, 6-12 hours, 12-24 hours, 24-48 hours

Additionally, patient demographics and clinical characteristics such as age, gender, BMI, and previous medical and surgical history will be collected. Procedural characteristics such as location of tracts (supracostal vs infracostal), size of nephrostomy tract, and type of nephrostomy tube will be recorded.

A secondary outcome that deserves further mention will be the total dose of narcotics from over the inpatient hospital course. This will be measured from 1 hour after the patient reaches the post-anesthesia care unit (PACU) until the discharge order is placed. All opiate medication will be converted morphine equivalents and the values will be reported as total number of milligrams of morphine. In order to help reduce variability due to variations in prescriber patterns, patients will be started on a pain regimen as followed.

Mild pain: 1 tablet PO Oxycodone 5mg/Acetaminophen 325mg q4 hours Moderate pain: 2 tablets PO Oxycodone 5mg/Acetaminophen 325mg q4 hours Severe pain: 1 mg IV hydromorphone q4 hours Breakthrough pain: 0.5 mg IV hydromorphone q4 hours The analgesic regimen can be altered by the physician or physician assistant treating the patient at their discretion but efforts will be maintained to follow this analgesic regimen. Amount of narcotics used will be gleaned from the electronic medical record upon discharge of the patient. Time to start recording analgesics will begin one hour after patient is sent to the PACU. This will help decrease variability in anesthesiologist and peri-anesthesia prescribing patterns immediately at the conclusion of the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18 years old
2. Patients with calculus disease that can be treated with PCNL

Exclusion Criteria:

1. Patients <18 years old.
2. Patients who are not able to give consent for study
3. Patients with active urinary tract infection
4. Pregnant women
5. Patients with hepatic insufficiency
6. Patients with more than 2 access tracts created
7. Allergies to bupivacaine or liposomal bupivacaine
8. Patients with chronic pain syndromes as determined by using >30mg oral morphine equivalents per day
9. Patients who are neurologically impaired and may have altered pain sensation due to previous diseases (e.g. paraplegics, quadriplegics, systemic neurological condition, etc.)
10. Patients who are undergoing staged procedures during that same hospital stay
11. Patients who are placed on patient controlled analgesia or patient controlled epidural analgesia
12. Patients who remain intubated after surgery
13. Patients who will have ureteral stents
14. Patients who do not require care in the intensive care unit
15. Patients who are mentally impaired.
16. Patients who are criminal prisoners.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Scores from the Visual Analog Scale for pain 24 hours post-procedurally in the liposomal bupivacaine group and the bupivacaine group | 24 hours
  Scores from the Visual Analog Scale for pain 24 hours post-procedurally in the liposomal bupivacaine group and the bupivacaine group

SECONDARY OUTCOMES:
narcotic usage | pain scores at 6, 12, 24, and 48 hours
  quantify mg of morphine equivalent used post operative

CONTACTS AND LOCATIONS:
Overall Officials: David M Hoenig, md, Principal Investigator — Urologist
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jonnavithula N, Pisapati MV, Durga P, Krishnamurthy V, Chilumu R, Reddy B. Efficacy of peritubal local anesthetic infiltration in alleviating postoperative pain in percutaneous nephrolithotomy. J Endourol. 2009 May;23(5):857-60. doi: 10.1089/end.2008.0634. PMID 19397429
- [Background] Lojanapiwat B, Chureemas T, Kittirattarakarn P. The efficacy of peritubal analgesic infiltration in postoperative pain following percutaneous nephrolithotomy - A prospective randomized controlled study. Int Braz J Urol. 2015 Sep-Oct;41(5):945-52. doi: 10.1590/S1677-5538.IBJU.2014.0471. PMID 26689520
- [Background] Cherian JJ, Barrington J, Elmallah RK, Chughtai M, Mistry JB, Mont MA. Liposomal Bupivacaine Suspension, Can Reduce Length of Stay and Improve Discharge Status of Patients Undergoing Total Hip Arthroplasty. Surg Technol Int. 2015 Nov;27:235-9. PMID 26680403
- [Background] Marcet JE, Nfonsam VN, Larach S. An extended paIn relief trial utilizing the infiltration of a long-acting Multivesicular liPosome foRmulation Of bupiVacaine, EXPAREL (IMPROVE): a Phase IV health economic trial in adult patients undergoing ileostomy reversal. J Pain Res. 2013 Jul 18;6:549-55. doi: 10.2147/JPR.S46467. Print 2013. PMID 23901290
- [Background] Vogel JD. Liposome bupivacaine (EXPAREL(R)) for extended pain relief in patients undergoing ileostomy reversal at a single institution with a fast-track discharge protocol: an IMPROVE Phase IV health economics trial. J Pain Res. 2013 Jul 29;6:605-10. doi: 10.2147/JPR.S46950. Print 2013. PMID 23935387
- [Background] Hu D, Onel E, Singla N, Kramer WG, Hadzic A. Pharmacokinetic profile of liposome bupivacaine injection following a single administration at the surgical site. Clin Drug Investig. 2013 Feb;33(2):109-15. doi: 10.1007/s40261-012-0043-z. PMID 23229686